CLINICAL TRIAL: NCT06409559
Title: A Randomized Prospective Study Comparing Rim Plate to Buttress Plate for Posterior Wall Acetabular Fractures With and Without Inter-fragmentary Screws
Brief Title: Rim Plate to Buttress Plate for Posterior Wall Acetabular Fractures With and Without Inter-fragmentary Screws
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, H. Claude Sagi, MD, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OS22025
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Acetabular Fracture

STUDY DESIGN:
Intervention Model Description: Parallel assignment to two different methods of screw and plate fixation of posterior wall acetabulum fractures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Rim plate group (Other): This group will consist of patients where the posterior wall fracture will be operatively stabilized with a pelvic reconstruction plate and interfragmentary screws placed through the plate.
  Interventions: Device: Pelvic reconstruction plate without interfragmentary screws
- Buttress plate group (Other): This group will consist of patients where the posterior wall fracture will be operatively fixed with a buttress plate applied under compression without interfragmentary lag or position screws.
  Interventions: Device: Pelvic reconstruction plate with interfragmentary screws

INTERVENTIONS:
Device: Pelvic reconstruction plate without interfragmentary screws — The posterior wall fracture will be operatively stabilized with a pelvic reconstruction plate and interfragmentary screws placed through the plate.
  Arms: Rim plate group
Device: Pelvic reconstruction plate with interfragmentary screws — The posterior wall fracture will be operatively fixed with a buttress plate applied under compression without interfragmentary lag or position screws.
  Arms: Buttress plate group

SUMMARY:
The hypothesis of this study is that the Rim Plate method utilizing interfragmentary screws placed through the plate will result in superior fixation, a lower rate of loss of reduction of the fracture fragment, better anatomic healing of the articular (joint) surface, a decreased rate of early post-traumatic arthritic changes of the joint (cartilage) surface, and improved functional outcomes.

DETAILED DESCRIPTION:
Study type: Interventional Estimated enrollment: 60 Allocation: block randomization. The block randomization method is designed to randomize subjects into groups that result in equal sample sizes. This method is used to ensure a balance in sample size across groups over time.

Interventional model: parallel assignment Description: two different methods of screw and plate fixation of posterior wall acetabulum fractures.

Time perspective: Prospective

Population:

Skeletally mature patients who have presented with an acute traumatic fracture of the posterior wall of acetabulum due to dislocation of the femoral head will be included in this study. All surgeons on the study routinely perform both types of repairs.

Treatment arms and Intervention:

Arm A: Rim plate group - This group will consist of 30 patients where the posterior wall fracture will be operatively stabilized with a pelvic reconstruction plate and interfragmentary screws placed through the plate.

Arm B: Buttress plate group - This group will consist of 30 patients where the posterior wall fracture will be operatively fixed with a buttress plate applied under compression without interfragmentary lag or position screws.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature males and females, ≥ 18 years old and with age less than 65 years.
2. Fracture of the acetabular posterior wall fracture due to acute traumatic hip dislocation, confirmed with anteroposterior pelvic or hip radiographs, and CT scan
3. Operative fixation of fractures within 14 days of presenting to the emergency room.
4. Patient was ambulatory prior to fracture, with or without walking aids
5. Medically optimized for operative intervention
6. Provision of informed consent by patient or legal guardian.

Exclusion Criteria:

1. Patients not suitable for internal fixation (severe osteoarthritis, rheumatoid arthritis, or pathologic fracture).
2. Pre-existing orthopedic fixation, implant, or prosthesis around the affected acetabulum.
3. Patients with metabolic bone disease including diagnosis of osteoporosis.
4. Patients with bony or soft tissue infections around the acetabulum.
5. Patients unable to provide informed consent.
6. Patients having other fractures of Pelvis or acetabulum other than an isolated posterior acetabular wall fracture.
7. Patients with previous history of acetabular fracture (operative or nonoperative)
8. Patients with previous history of hip pathology such as avascular necrosis, hip dysplasia, Legg-Calve Perthes Disease, or advanced degenerative arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Displacement of posterior wall acetabular fragment | 12 months
  Measured on immediate post-op CT and compared to measurement one year post-op
Healing of the posterior wall fragment | 12 months
  Measured on immediate post-op CT and compared to measurement one year post-op
Articular space loss | 12 months
  Degree and extent of articular space loss (chondrolysis)

SECONDARY OUTCOMES:
Modified Merle d'Aubigne score | 12 months
  Evaluates pain, gait and mobility
IOWA hip score | 12 months
  Hip rating system
PROMIS-10 score | 12 months
  A system of highly reliable, precise measures of patient-reported health status for physical, mental, and social well-being
SMFA score | 12 months
  Measure the functional status of patients with a broad range of musculoskeletal injuries and disorders
SF 36 score | 12 months
  Quantifies health status and measures health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati College of Medicine, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] JUDET R, JUDET J, LETOURNEL E. FRACTURES OF THE ACETABULUM: CLASSIFICATION AND SURGICAL APPROACHES FOR OPEN REDUCTION. PRELIMINARY REPORT. J Bone Joint Surg Am. 1964 Dec;46:1615-46. No abstract available. PMID 14239854
- [Background] Matta JM. Fractures of the acetabulum: accuracy of reduction and clinical results in patients managed operatively within three weeks after the injury. J Bone Joint Surg Am. 1996 Nov;78(11):1632-45. PMID 8934477
- [Background] Moed BR, Kregor PJ, Reilly MC, Stover MD, Vrahas MS. Current management of posterior wall fractures of the acetabulum. Instr Course Lect. 2015;64:139-59. PMID 25745901
- [Background] Pease F, Ward AJ, Stevenson AJ, Cunningham JL, Sabri O, Acharya M, Chesser T. Posterior wall acetabular fracture fixation: A mechanical analysis of fixation methods. J Orthop Surg (Hong Kong). 2019 Sep-Dec;27(3):2309499019859838. doi: 10.1177/2309499019859838. PMID 31311424
- [Background] Baumgaertner MR. Fractures of the posterior wall of the acetabulum. J Am Acad Orthop Surg. 1999 Jan;7(1):54-65. doi: 10.5435/00124635-199901000-00006. PMID 9916185
- [Background] D'AUBIGNE RM, POSTEL M. Functional results of hip arthroplasty with acrylic prosthesis. J Bone Joint Surg Am. 1954 Jun;36-A(3):451-75. No abstract available. PMID 13163078
- [Background] Larson CB. Rating scale for hip disabilities. Clin Orthop Relat Res. 1963;31:85-93. No abstract available. PMID 5888865
- [Background] Reeve BB, Hays RD, Bjorner JB, Cook KF, Crane PK, Teresi JA, Thissen D, Revicki DA, Weiss DJ, Hambleton RK, Liu H, Gershon R, Reise SP, Lai JS, Cella D; PROMIS Cooperative Group. Psychometric evaluation and calibration of health-related quality of life item banks: plans for the Patient-Reported Outcomes Measurement Information System (PROMIS). Med Care. 2007 May;45(5 Suppl 1):S22-31. doi: 10.1097/01.mlr.0000250483.85507.04. PMID 17443115
- [Background] Swiontkowski MF, Engelberg R, Martin DP, Agel J. Short musculoskeletal function assessment questionnaire: validity, reliability, and responsiveness. J Bone Joint Surg Am. 1999 Sep;81(9):1245-60. doi: 10.2106/00004623-199909000-00006. PMID 10505521
- [Background] Laucis NC, Hays RD, Bhattacharyya T. Scoring the SF-36 in Orthopaedics: A Brief Guide. J Bone Joint Surg Am. 2015 Oct 7;97(19):1628-34. doi: 10.2106/JBJS.O.00030. PMID 26446970